CLINICAL TRIAL: NCT00554151
Title: Mitral Adjustable Annuloplasty Ring Feasibility and Safety Study (MAARS) for Treatment of Patients With Mitral Valve Regurgitation in Open Surgical Repair
Brief Title: Mitral Adjustable Annuloplasty Ring Feasibility and Safety Study
Acronym: MAARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Vicki Bebeau, St. Jude Medical, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAARS CIP Version 5
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Adjustable Annuloplasty Ring — The investigational device is intended for use in the treatment of mitral valve regurgitation.

SUMMARY:
Evaluation of the technical feasibility and safety of the Mitral Adjustable Annuloplasty Ring.

DETAILED DESCRIPTION:
Establish the technical feasibility and safety of implantation of the investigation device, adjustment of the investigational device post-implantation, and the ability of the investigational device to reduce mitral valve regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged greater or equal to 18 to less than or equal to age 75.
* Patients with indications to undergo mitral valve repair consistent with ACC/AHA recommendations; including greater or equal to 2+ regurgitation by pre-operative TEE or TTE assessment.
* Candidate for cardiopulmonary bypass.
* A Left Ventricular Ejection Fraction greater or equal to 40%.
* Able and willing to comply with all study requirements, including the required study follow-up visits.
* Able and willing to five consent and follow study instructions.
* Female patients of childbearing potential (not surgically sterilized or more than one year postmenopausal), with a negative pregnancy test (serum beta-hCG) within 24 hours prior to mitral valve surgery.

Exclusion Criteria:

* Any previous cardiac surgery.
* Any interventional cardiology procedure within six months prior to study to include all patients that have had a drug eluting stent (DES) implanted within 6 months.
* Evidence of an acute Myocardial Infarction (MI) within 7 days of the intended treatment with the investigational device.
* Prior mitral valve surgery or valvuloplasty or currently implanted prosthetic valve.
* Restricted mobility of the mitral apparatus that results in a valvular area less than 3.0 cm2.
* Recent or evolving bacterial endocarditis or patients under current antibiotic therapy.
* Patients with ICD's.
* Any angiographic or clinical evidence that the investigator feels would place the patient at increased risk with the placement of the device or concurrent medical condition with a life expectancy of less than 12 months.
* Patients who are immunocompromised or with autoimmune diseases.
* Patients suffering from renal insufficiency (Creatinine >2.5 mg/dL) or patients with chronic renal failure undergoing dialysis.
* Co-morbid conditions that place the subject at an unacceptable surgical risk (e.g. sever chronic obstructive pulmonary disease, hepatic failure, immunosuppressive abnormalities, haematological abnormalities).
* Significant mitral annular calcification.
* Use of Coumadin, IIbIIIa inhibitors, Clopidigrel (Plavix) or other anti-coagulants within (5) five days prior to surgery.
* Participation in any study involving an investigational drug or device within the past month, or ongoing participation in a study with an investigational device.
* Intolerance or hypersensitivity to anaesthetics.
* Patients in whom transesophageal echo/Doppler is contraindicated.
* History of bleeding diathesis or coagulopathy.
* History of stroke within the prior 6 months
* Subjects to undergo concomitant cardiac repair or replacement other than CABG (less than or equal to 3 vessels) mitral annuloplasty, tricuspid valve repair and ablation therapy for correction of atrial fibrillation. Excluded concomitant procedures are: aortic valve replacement, LV remodeling, surgery and congenital repair.
* Patients with Euroscore > 10.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety: Freedom from major adverse events (MAE)at 30 days. Performance: Technical success rate of implantation of the investigation device. | 30 days, 90 days, 6 months and 1 year

SECONDARY OUTCOMES:
Ability to adjust the investigational device post-ring implantation after the patient has been weaned from CPB. MR reduction to <2+ post procedure, at post operative hospital discharge, at 30 days, at 6 months and one year. | 30 days, 90 days, 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: A. Franka Borger, Prof. MD, Principal Investigator — University Leipzig Germany; A.P. Kappetein, Dr., Principal Investigator — Erasmus MC, Universitair Medisch Centrum Rotterdam; R.J.M. Klautz, Dr., Principal Investigator — Leids Universitair Medisch Centrum Lieden; Anno Diegeler, Prof, MD, Principal Investigator — Herz-und Gefäß-Klinik GmbH Bad Neustadt; Ottavio Alfieri, Prof, MD, Principal Investigator — Hospital San Rafaele
Locations (5):
- Germany (2):
  - Herz - und Gefäß-Klinik GmbH Bad Neustadt, Bad Neustadt an der Saale, Saale
  - University Leipzig, Leipzig
- Hospital San Raffaele, Milan, Italy
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus MC, Universitair Medisch Centrum Rotterdam, Rotterdam